CLINICAL TRIAL: NCT06565442
Title: Feasibility of Using NeuraSignal Transcranial Doppler Robot for Generating Cerebral Autoregulation Curves in Neuro ICU Patients Admitted for Blood Pressure Management After Spinal Surgery
Brief Title: Feasibility of Using NeuraSignal Transcranial Doppler Robot
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Emily Wasson, MD, MPH Assistant Professor Division of Critical Care Department of Anesthesiology and Perioperative Medicine, University of Alabama at Birmingham
Other Study IDs: IRB-300013270; UAB (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2024-07-23; First posted 2024-08-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Autoregulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Group: Using the NeuraSignal transcranial doppler robot in a neuro ICU setting to measure cerebral blood flow correlated with arterial blood pressure to generate individualized cerebral autoregulatory curves.
  Interventions: Device: NeuraSignal transcranial doppler robot

INTERVENTIONS:
Device: NeuraSignal transcranial doppler robot — measure cerebral blood flow correlated with arterial blood pressure to generate individualized cerebral autoregulatory curves

SUMMARY:
The purpose of this study is to determine the feasibility of using the NeuraSignal transcranial doppler robot in a neuro ICU setting to measure cerebral blood flow correlated with arterial blood pressure to generate individualized cerebral autoregulatory curves

DETAILED DESCRIPTION:
This study aims to explore the feasibility of using the NeuraSignal transcranial doppler robot to generate cerebral autoregulation curves in adult patients admitted to the neuro ICU with a newly diagnosed brain mass. Cerebral blood flow measurements as calculated by a transcranial doppler robot will be time-correlated with arterial blood pressure measurements to generate personalized cerebral autoregulation curves. The study will be conducted prospectively and observationally on 20 patients as a pilot study for feasibility management.

Cerebral autoregulation has historically been difficult to quantify, in part due to the difficulty in measuring cerebral blood flow directly. Transcranial doppler (TCD) is a well-established method of calculating cerebral blood flow based on velocity through the middle cerebral arteries, however traditional methods of performing TCD are time consuming and require technical and procedural training. It also carries the established risk of miscalculation with variation in intra-operator technique differences and miscalculations due to inappropriate angle of the probe. The NeuraSignal transcranial doppler robot offers a potential tool to make obtaining cerebral blood flow calculations easier and, with the use of AI to determine optimal windows, significantly decreases intra-operator differences and errors associated with inappropriate probe angle. Cerebral blood flow calculated in this way can then be correlated with arterial blood pressure and used to build cerebral autoregulatory curves in near real time. This study aims to build on previous studies deriving and using personalized cerebral autoregulatory curves and determine the feasibility of using the TCD robot in this way to make individualized cerebral autoregulatory curves more accessible as a tool for personalized blood pressure management.

ELIGIBILITY:
Inclusion Criteria:

* 18-89
* Patients admitted to the Neuro ICU for blood pressure management (MAP management) after spinal surgery

Exclusion Criteria:

* Patients under 18 years (or bodyweight <50kg if age unknown),
* prisoners
* pregnant women,
* non-English speaking,
* patients enrolled in concurrent
* ongoing interventional trial
* students of UAB
* employees of UAB
* targeting specific populations
* patients with previously diagnosed brain pathology
* patients with open wounds over temporal bones precluding transcranial doppler

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Neuro ICU for blood pressure management (MAP management) after spinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-14 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | one year
  Cerebral autoregulatory curve generation using the NeuraSignal transcranial doppler robot correlated with arterial blood pressure measurements in neuro ICU patients admitted for blood pressure management after spinal surgery

SECONDARY OUTCOMES:
Secondary outcome | one year
  left or right shifting of the autoregulatory curve as a result of vasopressor use

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Wasson, MD,MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined.